CLINICAL TRIAL: NCT02661126
Title: A Two-Part, Open-Label Study to Investigate the Single-Dose Pharmacokinetics of MK-3682B (MK-3682/MK-5172/MK-8408 Fixed Dose Combination) When Administered to Subjects With Moderate and Severe Renal Insufficiency
Brief Title: Pharmacokinetics of MK-3682B in Participants With Moderate to Severe Renal Insufficiency (MK-3682B-030)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3682B-030; MK-3682B-030 (Other: Merck Protocol Number); CA16919 (Other: Celerion Protocol Number)
Record Dates: First submitted 2016-01-19; First posted 2016-01-22 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Moderate RI Participants (Experimental): Participants with an estimated glomerular filtration rate (eGFR) of ≥30 mL/min/1.73m^2 to <60 mL/min/1.73m^2 take 2 MK-3682B FDC tablets on Day 1 after fasting for 10 hours.
  Interventions: Drug: MK-3682B
- Severe RI Participants (Experimental): Participants with an eGFR of ≥15 mL/min/1.73m^2 to <30 mL/min/1.73m^2 take 2 MK-3682B FDC tablets on Day 1 after fasting for 10 hours.
  Interventions: Drug: MK-3682B
- Healthy Participants (Experimental): Healthy participants (creatinine clearance [CLcr] ≥80 mL/min) take 2 MK-362B FDC tablets on Day 1 after fasting for 10 hours. Healthy participants are matched to RI participants based on mean age, body mass index (BMI) and gender.
  Interventions: Drug: MK-3682B

INTERVENTIONS:
Drug: MK-3682B — FDC oral tablet containing 225 mg uprifosbuvir + 50 mg grazoprevir + 30 mg ruzasvir.

SUMMARY:
The purpose of this study is to compare the plasma pharmacokinetics (PK) of single doses of MK-3682B, a fixed dose combination (FDC) tablet containing uprifosbuvir (MK-3682) + grazoprevir (MK-5172) + ruzasvir (MK-8408) in participants with moderate (Part 1) and severe (Part 2) renal insufficiency (RI) to plasma PK in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Healthy adult males or females 18-80 years of age at screening
* Continuous non-smokers or moderate smokers (≤ 20 cigarettes/day or the equivalent) and agrees to consume no more than 10 cigarettes per day during the study period
* BMI ≥ 18 and ≤ 40.0 kg/m^2
* Agrees not to become pregnant or father a child during participation in the study
* Females of childbearing potential must either be abstinent for 14 days prior to dosing and throughout the study or be using an acceptable birth control method
* Vasectomized or non-vasectomized males must agree to use a condom with spermicide or abstain from sexual intercourse from the first dose until 90 days after dosing
* Males must agree not to donate sperm from dosing until 90 days after dosing

Moderate and Severe RI Participants:

* Baseline health is judged to be stable based on medical history, physical examination, laboratory profiles, vital signs, or electrocardiograms (ECGs), as deemed by the Investigator
* Has had no clinically significant change in renal status at least 1 month prior to dosing and is not currently or has not previously been on hemodialysis
* Moderate RI: has baseline eGFR ≥ 30 mL/min/1.73m^2 and < 60 mL/min/1.73m^2, based on the Modification of Diet in Renal Disease (MDRD) equation at screening
* Severe RI: has baseline eGFR ≥ 15 mL/min/1.73m^2 and < 30 mL/min/1.73m^2, based on the MDRD equation at screening

Healthy Participants:

* Is within ± 10 years of the mean age of moderate and severe RI arms
* BMI is within 10% of the mean BMI of participants with moderate and severe RI arms
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or ECGs, as deemed by the Investigator
* Baseline CLcr ≥ 80 mL/min based on Cockcroft-Gault equation at screening

Exclusion Criteria:

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator
* History of any illness that, in the opinion of the Investigator, might confound the results of the study or poses an additional risk by participating in the study
* Is female and pregnant or lactating
* Positive results for the urine or saliva drug screen or urine or breath alcohol screen at screening or check-in unless the positive drug screen is due to prescription drug use that is approved by the Investigator and Sponsor
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV)
* Seated heart rate is equal to or lower than 44 beats per minute (bpm) or higher than 100 bpm at screening
* Has had a renal transplant or has had nephrectomy
* Donation of blood or had significant blood loss within 56 days prior to dosing of study drug, or donation of plasma within 7 days prior to dosing
* Has participated in another clinical trial within 28 days prior to dosing of study drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2016-08-26 (Actual); Study Completion 2016-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Part 1, adults with moderate renal impairment (RI; determined by estimated glomerular filtration rate [eGFR]), and healthy participants, were recruited at 2 sites in the US. Part 2 was intended to enroll severe RI participants but was not conducted based on results of a planned interim analysis of Part 1 data.
Groups:
- Moderate RI Participants: Participants with an eGFR of ≥30 mL/min/1.73m^2 to <60 mL/min/1.73m^2 took 2 MK-3682B fixed dose combination (FDC) tablets (225 mg uprifosbuvir + 50 mg grazoprevir + 30 mg ruzasvir per tablet) on Day 1 after fasting for 10 hours.
- Healthy Participants: Healthy participants (creatinine clearance [CLcr] ≥80 mL/min) took 2 MK-362B FDC tablets (225 mg uprifosbuvir + 50 mg grazoprevir + 30 mg ruzasvir per tablet) on Day 1 after fasting for 10 hours.
Period: Overall Study
Arm/Group | Moderate RI Participants | Healthy Participants
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Moderate RI Participants: Participants with an eGFR of ≥30 mL/min/1.73m^2 to <60 mL/min/1.73m^2 took 2 MK-3682B FDC tablets (225 mg uprifosbuvir + 50 mg grazoprevir + 30 mg ruzasvir per tablet) on Day 1 after fasting for 10 hours.
- Healthy Participants: Healthy participants (CLcr ≥80 mL/min) took 2 MK-362B FDC tablets (225 mg uprifosbuvir + 50 mg grazoprevir + 30 mg ruzasvir per tablet) on Day 1 after fasting for 10 hours.
- Total: Total of all reporting groups
Arm/Group | Moderate RI Participants | Healthy Participants | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] — Healthy participants were matched to moderate RI participants based on age.
  Years | 69.6 (9.0) | 65.8 (2.6) | 67.7 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Healthy participants were matched to moderate RI participants based on gender.
  Participants
    Female | 2 | 2 | 4
    Male | 6 | 6 | 12
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Healthy participants were matched to moderate RI participants based on BMI.
  kg/m^2 | 30.32 (4.023) | 30.11 (2.057) | 30.22 (3.088)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Dosing to Time of Last Measurable Concentration (AUC0-last) of Uprifosbuvir (MK-3682)
Description: AUC0-last is a measure of total exposure to uprifosbuvir in plasma from the start of dosing to the time of the last quantifiable (< lower limit of quantification [LLOQ]) sample following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
uM*hr | 8.55 [6.22 to 11.8] | 4.23 [3.08 to 5.82]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — Geometric least-squares mean ratio (GMR) of AUC0-last in Moderate RI/Healthy Participants; GMR of AUC0-last in Moderate RI/Healthy = 2.02, 90% CI 2-sided [1.40 to 2.92]

2. Primary Outcome: AUC From Dosing to Infinity (AUC0-∞) of Uprifosbuvir
Description: AUC0-∞ is a measure of total exposure to uprifosbuvir in plasma from the start of dosing to infinity following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
uM*hr | 8.56 [6.24 to 11.7] | 4.28 [3.12 to 5.87]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of AUC0-∞ in Moderate RI/Healthy Participants; GMR of AUC0-∞ in Moderate RI/Healthy = 2.00, 90% CI 2-sided [1.39 to 2.89]

3. Primary Outcome: AUC From Dosing to 24 Hours Post-dose (AUC0-24) of Uprifosbuvir
Description: AUC0-24 is a measure of total exposure to uprifosbuvir in plasma from dosing to 24 hours following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, and 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
uM*hr | 8.54 [6.22 to 11.7] | 4.24 [3.08 to 5.82]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of AUC0-24 in Moderate RI/Healthy Participants; GMR of AUC0-24 in Moderate RI/Healthy = 2.02, 90% CI 2-sided [1.39 to 2.92]

4. Primary Outcome: Maximum Plasma Concentration (Cmax) of Uprifosbuvir
Description: Cmax is the maximum amount of uprifosbuvir in plasma following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
nM | 3030 [2230 to 4110] | 1570 [1160 to 2130]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of Cmax in Moderate RI/Healthy Participants; GMR of Cmax in Moderate RI/Healthy = 1.92, 90% CI 2-sided [1.35 to 2.74]

5. Primary Outcome: Plasma Concentration 24 Hours Post-dose (C24) of Uprifosbuvir
Description: C24 is the plasma concentration of uprifosbuvir 24 hours following oral administration of MK-3682B.
Time Frame: 24 hours post-dose
Population: All Healthy Control participants are included in the analysis. Since >50% of participants in the Moderate RI group had C24 values <LLOQ, no data are presented for this group as per Merck policy.
Measure: Median (Full Range); unit: nM
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 0 | 8
nM |  | 3.65 [0.00 to 9.97]

6. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Uprifosbuvir
Description: Tmax is the time required to reach the maximum post-dose plasma concentration of uprifosbuvir following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis
Measure: Median (Full Range); unit: Hours
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
Hours | 1.00 [0.50 to 4.00] | 1.00 [0.50 to 2.00]

7. Primary Outcome: Apparent Total Body Clearance (CL/F) of Uprifosbuvir
Description: CL/F is the apparent total body clearance of uprifosbuvir following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
Liters/hour | 96.3 (51.5) | 193 (34.7)

8. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Uprifosbuvir
Description: Vz/F is the apparent volume of distribution of uprifosbuvir following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
Liters | 290 (51.7) | 724 (115.2)

9. Primary Outcome: Apparent Terminal Half-life in Plasma (t½) of Uprifosbuvir
Description: t1/2 is the amount of time required to clear 50% of uprifosbuvir from plasma following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
Hours | 2.09 (65.6) | 2.60 (92.9)

10. Primary Outcome: AUC0-last of Uprifosbuvir Metabolite M5
Description: AUC0-last is a measure of total exposure to uprifosbuvir metabolite M5 in plasma from the start of dosing to the time of the last quantifiable (<LLOQ) sample following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
uM*hr | 14.8 [11.1 to 19.6] | 7.62 [5.74 to 10.1]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of AUC0-last in Moderate RI/Healthy Participants; GMR of AUC0-last in Moderate RI/Healthy = 1.94, 90% CI 2-sided [1.39 to 2.72]

11. Primary Outcome: AUC0-∞ of Uprifosbuvir Metabolite M5
Description: AUC0-∞ is a measure of total exposure to uprifosbuvir metabolite M5 in plasma from the start of dosing to infinity following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
uM*hr | 16.2 [12.5 to 20.8] | 7.99 [6.19 to 10.3]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of AUC0-∞ in Moderate RI/Healthy Participants; GMR of AUC0-∞ in Moderate RI/Healthy = 2.02, 90% CI 2-sided [1.50 to 2.74]

12. Primary Outcome: AUC0-24 of Uprifosbuvir Metabolite M5
Description: AUC0-24 is a measure of total exposure to uprifosbuvir metabolite M5 in plasma from dosing to 24 hours following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, and 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
uM*hr | 4.59 [3.25 to 6.47] | 2.67 [1.89 to 3.77]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of AUC0-24 in Moderate RI/Healthy Participants; GMR of AUC0-24 in Moderate RI/Healthy = 1.72, 90% CI 2-sided [1.15 to 2.56]

13. Primary Outcome: Cmax of Uprifosbuvir Metabolite M5
Description: Cmax is the maximum amount of uprifosbuvir metabolite M5 in plasma following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
nM | 321 [220 to 467] | 173 [119 to 252]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of Cmax in Moderate RI/Healthy Participants; GMR of Cmax in Moderate RI/Healthy = 1.85, 90% CI 2-sided [1.20 to 2.87]

14. Primary Outcome: C24 of Uprifosbuvir Metabolite M5
Description: C24 is the plasma concentration of uprifosbuvir metabolite M5 24 hours following oral administration of MK-3682B.
Time Frame: 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
nM | 262 [189 to 365] | 129 [93.0 to 180]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of C24 in Moderate RI/Healthy Participants; GMR of C24 in Moderate RI/Healthy = 2.03, 90% CI 2-sided [1.38 to 2.97]

15. Primary Outcome: Tmax of Uprifosbuvir Metabolite M5
Description: Tmax is the time required to reach the maximum post-dose plasma concentration of uprifosbuvir metabolite M5 following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis
Measure: Median (Full Range); unit: Hours
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
Hours | 20.00 [10.00 to 24.00] | 13.00 [12.00 to 16.00]

16. Primary Outcome: Lag Time (Tlag) of Uprifosbuvir Metabolite M5
Description: Tlag is the time from dosing to first appearance in plasma of uprifosbuvir metabolite M5 following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis
Measure: Median (Full Range); unit: Hours
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
Hours | 2.00 [2.00 to 3.00] | 2.00 [2.00 to 3.00]

17. Primary Outcome: t½ of Uprifosbuvir Metabolite M5
Description: t1/2 is the amount of time required to clear 50% of uprifosbuvir metabolite M5 from plasma following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
Hours | 26.27 (45.0) | 25.33 (6.4)

18. Primary Outcome: AUC0-last of Uprifosbuvir Metabolite M6
Description: AUC0-last is a measure of total exposure to uprifosbuvir metabolite M6 in plasma from the start of dosing to the time of the last quantifiable (<LLOQ) sample following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
uM*hr | 63.9 [50.1 to 81.5] | 33.5 [26.3 to 42.8]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of AUC0-last in Moderate RI/Healthy Participants; GMR of AUC0-last in Moderate RI/Healthy = 1.91, 90% CI 2-sided [1.44 to 2.53]

19. Primary Outcome: AUC0-∞ of Uprifosbuvir Metabolite M6
Description: AUC0-∞ is a measure of total exposure to uprifosbuvir metabolite M6 in plasma from the start of dosing to infinity following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
uM*hr | 71.4 [55.8 to 91.3] | 36.2 [28.3 to 46.2]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of AUC0-∞ in Moderate RI/Healthy Participants; GMR of AUC0-∞ in Moderate RI/Healthy = 1.97, 90% CI 2-sided [1.48 to 2.63]

20. Primary Outcome: AUC0-24 of Uprifosbuvir Metabolite M6
Description: AUC0-24 is a measure of total exposure to uprifosbuvir metabolite M6 in plasma from dosing to 24 hours following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, and 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
uM*hr | 27.2 [22.2 to 33.4] | 13.9 [11.3 to 17.1]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of AUC0-24 in Moderate RI/Healthy Participants; GMR of AUC0-24 in Moderate RI/Healthy = 1.96, 90% CI 2-sided [1.54 to 2.48]

21. Primary Outcome: Cmax of Uprifosbuvir Metabolite M6
Description: Cmax is the maximum amount of uprifosbuvir metabolite M6 in plasma following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
nM | 1540 [1210 to 1950] | 906 [715 to 1150]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of Cmax in Moderate RI/Healthy Participants; GMR of Cmax in Moderate RI/Healthy = 1.70, 90% CI 2-sided [1.29 to 2.24]

22. Primary Outcome: C24 of Uprifosbuvir Metabolite M6
Description: C24 is the plasma concentration of uprifosbuvir metabolite M6 24 hours following oral administration of MK-3682B.
Time Frame: 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
nM | 905 [712 to 1150] | 466 [367 to 592]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of C24 in Moderate RI/Healthy Participants; GMR of C24 in Moderate RI/Healthy = 1.94, 90% CI 2-sided [1.47 to 2.57]

23. Primary Outcome: Tmax of Uprifosbuvir Metabolite M6
Description: Tmax is the time required to reach the maximum post-dose plasma concentration of uprifosbuvir metabolite M6 following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis
Measure: Median (Full Range); unit: Hours
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
Hours | 8.00 [3.00 to 10.00] | 3.50 [3.00 to 4.00]

24. Primary Outcome: t½ of Uprifosbuvir Metabolite M6
Description: t1/2 is the amount of time required to clear 50% of uprifosbuvir metabolite M6 from plasma following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
Hours | 33.58 (39.7) | 30.55 (19.7)

25. Primary Outcome: AUC0-last of Grazoprevir (MK-5172)
Description: AUC0-last is a measure of total exposure to grazoprevir in plasma from the start of dosing to the time of the last quantifiable (<LLOQ) sample following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
uM*hr | 0.974 [0.523 to 1.81] | 0.730 [0.392 to 1.36]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of AUC0-last in Moderate RI/Healthy Participants; GMR of AUC0-last in Moderate RI/Healthy = 1.33, 90% CI 2-sided [0.65 to 2.75]

26. Primary Outcome: AUC0-∞ of Grazoprevir
Description: AUC0-∞ is a measure of total exposure to grazoprevir in plasma from the start of dosing to infinity following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants except 1 are included in the analysis. One participant in the Moderate RI group did not have a well characterized terminal phase and their value was set to "missing".
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 7 | 8
uM*hr | 1.32 [0.708 to 2.45] | 0.826 [0.463 to 1.48]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of AUC0-∞ in Moderate RI/Healthy Participants; GMR of AUC0-∞ in Moderate RI/Healthy = 1.59, 90% CI 2-sided [0.79 to 3.19]

27. Primary Outcome: AUC0-24 of Grazoprevir
Description: AUC0-24 is a measure of total exposure to grazoprevir in plasma from the start of dosing to 24 hours post-dose following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, and 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
uM*hr | 0.436 [0.218 to 0.875] | 0.380 [0.190 to 0.762]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of AUC0-24 in Moderate RI/Healthy Participants; GMR of AUC0-24 in Moderate RI/Healthy = 1.15, 90% CI 2-sided [0.51 to 2.57]

28. Primary Outcome: Cmax of Grazoprevir
Description: Cmax is the maximum amount of grazoprevir in plasma following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
nM | 67.5 [31.0 to 147] | 54.7 [25.1 to 119]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of Cmax in Moderate RI/Healthy Participants; GMR of Cmax in Moderate RI/Healthy = 1.23, 90% CI 2-sided [0.50 to 3.05]

29. Primary Outcome: C24 of Grazoprevir
Description: C24 is the plasma concentration of grazoprevir 24 hours following oral administration of MK-3682B.
Time Frame: 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
nM | 9.41 [4.64 to 19.1] | 7.36 [3.63 to 14.9]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of C24 in Moderate RI/Healthy Participants; GMR of C24 in Moderate RI/Healthy = 1.28, 90% CI 2-sided [0.56 to 2.91]

30. Primary Outcome: Tmax of Grazoprevir
Description: Tmax is the time required to reach the maximum post-dose plasma concentration of grazoprevir following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis
Measure: Median (Full Range); unit: Hours
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
Hours | 2.00 [1.00 to 4.00] | 2.25 [1.00 to 10.00]

31. Primary Outcome: CL/F of Grazoprevir
Description: CL/F is the apparent total body clearance of grazoprevir following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 7 | 8
Liters/hour | 99.1 (122.0) | 158 (57.9)

32. Primary Outcome: Vz/F of Grazoprevir
Description: Vz/F is the apparent volume of distribution of grazoprevir following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 7 | 8
Liters | 6030 (183.5) | 9750 (77.5)

33. Primary Outcome: t½ of Grazoprevir
Description: t1/2 is the amount of time required to clear 50% of grazoprevir from plasma following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 7 | 8
Hours | 42.21 (40.3) | 42.85 (26.4)

34. Primary Outcome: AUC0-last of Ruzasvir (MK-8408)
Description: AUC0-last is a measure of total exposure to ruzasvir in plasma from the start of dosing to the time of the last quantifiable (<LLOQ) sample following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
uM*hr | 2.07 [1.60 to 2.67] | 1.32 [1.03 to 1.71]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of AUC0-last in Moderate RI/Healthy Participants; GMR of AUC0-last in Moderate RI/Healthy = 1.56, 90% CI 2-sided [1.19 to 2.05]

35. Primary Outcome: AUC0-∞ of Ruzasvir
Description: AUC0-∞ is a measure of total exposure to ruzasvir in plasma from the start of dosing to infinity following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
uM*hr | 2.19 [1.71 to 2.81] | 1.40 [1.09 to 1.79]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of AUC0-∞ in Moderate RI/Healthy Participants; GMR of AUC0-∞ in Moderate RI/Healthy = 1.57, 90% CI 2-sided [1.20 to 2.05]

36. Primary Outcome: AUC0-24 of Ruzasvir
Description: AUC0-24 is a measure of total exposure to ruzasvir in plasma from dosing to 24 hours following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, and 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
uM*hr | 1.11 [0.872 to 1.42] | 0.744 [0.583 to 0.948]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of AUC0-24 in Moderate RI/Healthy Participants; GMR of AUC0-24 in Moderate RI/Healthy = 1.49, 90% CI 2-sided [1.13 to 1.98]

37. Primary Outcome: Cmax of Ruzasvir
Description: Cmax is the maximum amount of ruzasvir in plasma following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
nM | 117 [88.9 to 154] | 80.9 [61.6 to 106]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of Cmax in Moderate RI/Healthy Participants; GMR of Cmax in Moderate RI/Healthy = 1.44, 90% CI 2-sided [1.05 to 1.98]

38. Primary Outcome: C24 of Ruzasvir
Description: C24 is the plasma concentration of ruzasvir 24 hours following oral administration of MK-3682B.
Time Frame: 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
nM | 23.9 [18.5 to 30.8] | 15.5 [12.0 to 20.0]
Statistical Analysis 1: Comparison: Moderate RI Participants vs Healthy Participants; Test type: Other — GMR of C24 in Moderate RI/Healthy Participants; GMR of C24 in Moderate RI/Healthy = 1.54, 90% CI 2-sided [1.15 to 2.07]

39. Primary Outcome: Tmax of Ruzasvir
Description: Tmax is the time required to reach the maximum post-dose plasma concentration of ruzasvir following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis
Measure: Median (Full Range); unit: Hours
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
Hours | 3.00 [1.50 to 4.00] | 3.00 [2.00 to 4.00]

40. Primary Outcome: CL/F of Ruzasvir
Description: CL/F is the apparent total body clearance of ruzasvir following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
Liters/hour | 31.0 (34.5) | 48.8 (31.2)

41. Primary Outcome: Vz/F of Ruzasvir
Description: Vz/F is the apparent volume of distribution of ruzasvir following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
Liters | 1410 (40.0) | 2060 (26.9)

42. Primary Outcome: t½ of Ruzasvir
Description: t1/2 is the amount of time required to clear 50% of ruzasvir from plasma following oral administration of MK-3682B.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Moderate RI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8
Hours | 31.50 (11.4) | 29.31 (7.0)

ADVERSE EVENTS:
Time Frame: Up to 14 days
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. All 16 participants were included in the safety and tolerability assessment.
Arm/Group | Moderate RI Participants | Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate RI Participants (N=8) | Healthy Participants (N=8)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No